CLINICAL TRIAL: NCT02706106
Title: Assessment of a Knee Brace in Patients With Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Marco Aurélio Nemitalla Added, Master in Science, Irmandade da Santa Casa de Misericordia de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCMAA01
Record Dates: First submitted 2015-11-28; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Knee brace with a hole (Experimental): Patients will be prepared to receive the device of knee brace with a hole in the sit position. This intervention will be blinded. Patients will receive a mask covering their eyes and the knee brace will be placed by the researchers, then the knee area will be covered with a dark clothing bag, so the patient will not be able to guess which type of brace is wearing (with or without a hole). Patient will perform the tests without the mask covering their eyes and only the dark clot bag on their knee.
  Interventions: Device: Knee brace
- Knee brace without a hole (Placebo Comparator): Patients will be prepared to receive the device of knee brace without a hole in the sit position. This intervention will be blinded. Patients will receive a mask covering their eyes and the knee brace will be placed by the researchers, then the knee area will be covered with a dark clothing bag, so the patient will not be able to guess which type of brace is wearing (with or without a hole). Patient will perform the tests without the mask covering their eyes and only the dark clot bag on their knee.
  Interventions: Device: Knee brace

INTERVENTIONS:
Device: Knee brace — Patients will be prepared to receive the device of knee brace with or without a hole in the sit position. This intervention will be blinded. Patients will receive a mask covering their eyes and the knee brace will be placed by the researchers, then the knee area will be covered with a dark clothing bag, so the patient will not be able to guess which type of brace is wearing (with or without a hole). Patient will perform the tests without the mask covering their eyes and only the dark clot bag on their knee.

SUMMARY:
It is a controlled clinical trial randomized, double-blind evaluator. Will be considered eligible patients, individuals of both sexes, aged 40 -60, to submit at least four items of knee osteoarthrosis classification criteria, according to the American College of Rheumatology, pain above four points in the visual analogue scale (VAS), diagnosed with knee osteoarthritis and who sought physical therapy treatment.

Patients will be randomized by a number sequence generated by a computer using Microsoft Excel (Microsoft Corporation, Redmond, Washington), in opaque envelopes by researcher who will not attend the study.Patients will be divided into two groups: group with knee patellar hole or group without knee patellar hole. Shortly after the selection of the knee, the patient will have his eyes blind or cover in order to keep it '' blind '' regarding the type of knee brace that it would use.

Finally evaluator 1 will cover the knee with a black cloak, making the second evaluator ''blind '' regarding the type of knee brace that will be used.

Two investigators will carry out the data collection. The first evaluator will collect information on the clinical characteristics of patients, including evaluation form, numerical pain scale, which measures the intensity of pain, test Time Up and Go (TUG) test that measures the basic mobility of movement and test walking eight meters, whose purpose is to measure the time that the individual takes to walk a distance of eight meters.

ELIGIBILITY:
Inclusion Criteria:

* individuals of both sexes
* aged 40 -60
* at least four items of knee osteoarthrosis classification criteria, according to the American College of Rheumatology,
* pain above four points in the visual analogue scale (VAS)
* diagnosed with knee osteoarthritis
* no physical therapy treatment prior

Exclusion Criteria:

* neurological impairment
* partial or total knee prosthesis
* cardio-respiratory diseases
* pregnant women
* individuals who failed to perform the tests proposed

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change on pain sensation | Pain will be measured before and right after or maximum five minutes after wearing the brace knee
  Change on pain sensation will be compared from the baseline (before wearing the brace knee) with the pain sensation right after or maximum five minutes after wearing the brace knee. This evaluation will be performed asking the patient to identify their pain sensation by the visual analogue scale (VAS).

SECONDARY OUTCOMES:
Change on leg function | Leg function will be measured before and right after or maximum five minutes after wearing the brace knee
  Change on leg function will be measured before wearing the knee brace (baseline) and compared with right after or maximum five minutes after wearing the knee brace evaluation. Leg function will be assessed by Time Up and Go (TUG) test.
Change on agility | Agility will be measured before and right after or maximum five minutes after wearing the brace knee
  Change on agility will be measured before wearing the knee brace (baseline) and compared to right after or maximum five minutes after wearing the brace knee evaluation. Agility will be assessed by 8 Meter Walk test. The time to complete this test will be recorded by the researchers and this time will be the result considered for comparison from baseline and after wearing the knee brace.

CONTACTS AND LOCATIONS:
Overall Officials: Marco N Added, MSc, Principal Investigator — Irmandade da Santa Casa de Misericórdia de São Paulo
Locations (1):
- Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes